CLINICAL TRIAL: NCT05120154
Title: Improving Palliative Care in the Home and Community: Building CAPACITI (Community Access to Palliative Care Via Interprofessional Primary Care Teams Improvement) Cluster Randomized Controlled Trial
Brief Title: Building CAPACITI for Community-Based Palliative Care
Acronym: CAPACITI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 13867
Record Dates: First submitted 2021-10-15; First posted 2021-11-15 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Palliative Care
Keywords: Palliative care; CAPACITI; End of life; Primary care; Early identification
MeSH Terms: conditions — Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Access to all the CAPACITI module materials, provided on a learning management system. The intervention group will also receive the CAPACITI program with module facilitation, namely high-facilitation and expert coaching in the coverage of module materials in four live webinars (bimonthly for the 2 month duration of the module = 4 webinars).
  Interventions: Other: Online educational materials; Behavioral: Facilitated online webinars
- Control (Active Comparator): Access to all the CAPACITI module materials, provided on a learning management system. The control group will not receive module facilitation (i.e., will entail self-directed learning).
  Interventions: Other: Online educational materials

INTERVENTIONS:
Other: Online educational materials — The CAPACITI program is comprised of three independent modules, taken separately (each constituting an intervention): (1) Identify and Assess; (2) Enhance Communication Skills; (3) Enhance Skills for Ongoing Care (including involvement of family and specialists). Each module addresses a critical component of implementing a palliative care approach into primary care practice. The CAPACITI program emphasizes practice supports in each module, integrating two components: 1) clinical education in the form of expert advice and tips, and 2) evidence-based tools with action steps.
Behavioral: Facilitated online webinars — Intervention participants will be invited to participate in facilitated online discussions. These discussions review the online materials and share strategies for problem-solving.
  Arms: Intervention

SUMMARY:
The purpose of this cluster randomized controlled trial is to assess the efficacy of a quality improvement intervention called CAPACITI intended to increase competency among primary care teams to deliver early palliative care. CAPACITI is palliative care training and coaching program for primary care teams, comprised of three, two-month (4 session) modules, each addressing a critical component of implementing a palliative care approach into primary care practice.

DETAILED DESCRIPTION:
Improving access to home-based palliative care can improve patient and system outcomes; however, there is a lack of programs to build capacity among primary care teams to deliver this care. To address this gap, the investigators are offering a quality improvement intervention called CAPACITI. CAPACITI is palliative care training and coaching program for primary care teams, comprised of three, two-month (4 session) modules. Each module addresses a critical component of implementing a PC approach into primary care practice: (1) Identify and Assess; (2) Enhance Communication Skills; (3) Enhance Skills for Ongoing Care (including involvement of family and specialists). Over bi-monthly (one hour) sessions, each CAPACITI module uniquely integrates 3 components: clinical education in the form of expert advice and tips; evidence-based tools; and high-facilitation and expert coaching for adaptation to local context. The study will offer the CAPACITI modules to primary care teams across Canada. Teams that register for a module will be randomized to one of two arms: 1) facilitated learning where the module materials are covered in live webinars, and 2) non-facilitated learning where teams have access to all module materials to use a self-directed approach. The online materials for both study arms will be provided on a learning management system. The investigators will examine the difference between the facilitated and nonfacilitated approaches in teams' abilities to provide a palliative care approach in relation to the content of the module. Ultimately this research program will strengthen the primary care system and increase access to home-based palliative care for patients across Canada.

ELIGIBILITY:
Inclusion Criteria:

* Each team must be comprised of primary care providers, defined as having a minimum of at least 1 of the following: family physician, nurse practitioner, or nurse and practice coordinator (including manager or administrator) that provides primary care. Teams can be a single provider. Teams can also have other team members (e.g. social worker, pharmacist, etc.).
* Each team must be community-based and willing to provide palliative care, defined as managing symptoms, addressing psychosocial needs, educating patients and families, and coordinating care.

Exclusion Criteria:

* Not community-based
* Not willing to provide palliative care
* Outside of Canada

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Proportion of case load identified as requiring a palliative care approach | Up to one month post module
  Measured based on self-reported i) Number of patients in caseload and number (calculated %) reported as identified as requiring a palliative care approach, ii) Typical timing of when to initiate a palliative care approach for cancer and non-cancer patients respectively.
End-of-Life Professional Caregiver Survey (EPCS) | Up to one month post module
  The EPCS is a 28-item scale developed to assess palliative care-specific educational needs within an interprofessional team related to three main subdomains: Effective Care Delivery (ECD 8-items); Patient and Family-Centered Communication (PFCC 12-items); and Cultural and Ethical Values (CEV 8-items) (Lazenby, 2012). Each item is scored on a 5-point Likert scale ranging from 1 (lowest level of skill) to 5 (greatest level of skill). Items represent care-provider comfort with a variety of situations related to palliative and EOL care. The EPCS covers all eight domains of the national palliative care guidelines and core lessons of physician-specific and nurse-specific end of life education curricula in the USA. The EPCS exhibits strong internal consistency (alpha = 0.96). For the purposes of this study we will exclude the CEV sub-domain items from the EPCS.
Assignment Completion & Change Survey | Up to one month post module
  This survey is a two-part, study created questionnaire based on the CAPACITI module activities. Part A is unique to each module, asking participants to indicate the extent to which they were able to complete each of the session assignments for the module. Response options are: Have not started (1), Started but not completed (2), Completed (3). Part B contains four items assessing changes in thinking, behaviour, processes, and patient/family experience, respectively. Each item is scored on a 5-point Likert scale, rating the strength of agreement with each element of change, from 1 (strongly disagree) to 5 (strongly agree).

SECONDARY OUTCOMES:
CAPACITI Competencies Survey | Up to one month post module
  The CAPACITI Competencies Survey is a study created questionnaire based on the CanMEDS framework for improving patient care by enhancing physician training and the topics covered in the CAPACITI program. CanMEDS, developed by the Royal College of Physicians, delineates critical competencies to effectively meeting the health care needs of patients, including communication, expertise, collaboration, advocacy, and commitment (cite https://www.royalcollege.ca/rcsite/canmeds/canmeds-framework-e). Each item is scored on a 7-point Likert scale ranging from 1 (lowest level of confidence) to 7 (greatest level of confidence). The Competencies Survey was developed and tested in the CAPACITI pilot study. The CAPACITI Competencies Survey exhibits strong internal consistency (alpha = 0.96).
Assessment of Interprofessional Team Collaboration Scale II (AITCS II) | Up to one month post module
  The AITCS is an instrument designed to measure interprofessional collaboration among team members. The AITCS consists of 23 items considered characteristic of interprofessional collaboration (how team works and acts). Scale items represent three elements considered to be key to collaborative practice. These subscales are: Partnership (8 items), Cooperation (8 items), and Coordination (7 items). Each item is scored on a 5-point Likert scale indicating the extent to which the team exhibits each, ranging from 1 (Never) to 5 (Always). Internal consistency estimates for reliability of each subscale range from 0.80 to 0.97, with an overall reliability of 0.98.
Module Session Evaluation | Up to one month post module
  Participants will be asked to complete an evaluation poll at the end of each module session, consisting of 4 items: 3 items scored on a 5-point Likert scale ranging from 1 (Not at all/ Poor/ Not successful) to 5 (Very likely/ Excellent / Extremely successful) and 1 dichotomous item assessing perceived bias (Yes/No).

CONTACTS AND LOCATIONS:
Overall Officials: Hsien Seow, PhD, Principal Investigator — Department of Oncology, McMaster University and Juravinski Cancer Centre
Locations (1):
- Juravinski Cancer Centre - Hamilton Health Sciences, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Derived] Matthew M, Bainbridge D, Myers J, Levine O, Steinberg L, Incardona N, Winemaker S, Kortes-Miller K, Stajduhar K, Kilbertus F, Pereira J, Seow H. Facilitated Versus Self-Directed Educational Modalities in Palliative Care Training: A Randomized Controlled Trial of the CAPACITI Intervention. Palliat Med Rep. 2025 Jun 17;6(1):365-373. doi: 10.1089/pmr.2025.0010. eCollection 2025. PMID 40919547
- [Derived] Seow H, Bainbridge D, Winemaker S, Stajduhar K, Pond G, Kortes-Miller K, Marshall D, Kilbertus F, Myers J, Steinberg L, Incardona N, Levine O, Pereira J. Increasing palliative care capacity in primary care: study protocol of a cluster randomized controlled trial of the CAPACITI training program. BMC Palliat Care. 2023 Jan 5;22(1):2. doi: 10.1186/s12904-022-01124-x. PMID 36604714

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/54/NCT05120154/Prot_SAP_000.pdf